CLINICAL TRIAL: NCT05114863
Title: An In-Clinic Confinement Study to Assess Elements of Abuse Liability for a Heated Tobacco Product (20020064) With Four Non-Combusted Cigarette Variants (40007385 - 40007388)
Brief Title: CSD200907: A Study to Assess Elements of Abuse Liability for a Heated Tobacco Product With Four Non-Combusted Cigarette Variants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD200907
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-menthol smokers (Experimental): Subjects will be randomized to one of ten product use sequences, such that one of the five IPs (A1,B,C,D,N) will be used in each of the five Test Sessions.
  Interventions: Other: Product A1; Other: Product B; Other: Product C; Other: Product D; Other: Product N
- Menthol smokers (Experimental): Subjects will be randomized to one of six product use sequences, such that one of the six IPs (A2,E,F,G,H,N) will be used in each of the six Test Sessions.
  Interventions: Other: Product A2; Other: Product E; Other: Product F; Other: Product G; Other: Product H; Other: Product N

INTERVENTIONS:
Other: Product A1 — Usual Brand (UB) filtered, non-menthol cigarette
  Arms: Non-menthol smokers
Other: Product B — 40007388, A Non-Combusted Cigarette Variant and product use Mode A
  Arms: Non-menthol smokers
Other: Product C — 40007388, A Non-Combusted Cigarette Variant and product use Mode B
  Arms: Non-menthol smokers
Other: Product D — 40007386, A Non-Combusted Cigarette Variant and product use Mode B
  Arms: Non-menthol smokers
Other: Product A2 — Usual Brand (UB) filtered, menthol cigarette
  Arms: Menthol smokers
Other: Product E — 40007385, A Non-Combusted Cigarette Variant and product use Mode A
  Arms: Menthol smokers
Other: Product F — 40007385, A Non-Combusted Cigarette Variant and product use Mode B
  Arms: Menthol smokers
Other: Product G — 40007387, A Non-Combusted Cigarette Variant and product use Mode B
  Arms: Menthol smokers
Other: Product H — 40007386, A Non-Combusted Cigarette Variant and product use Mode B
  Arms: Menthol smokers
Other: Product N — Nicorette® White Ice Mint 4 mg nicotine gum

SUMMARY:
This is a single-center, open-label, randomized, 2-arm, within-arm cross-over study designed to evaluate elements of abuse liability (AL) including subjective effects and physiological measures (pharmacodynamics [PD]), and plasma nicotine uptake (pharmacokinetics [PK]) during and following ad libitum use of the study investigational products (IPs) by generally healthy smokers.

DETAILED DESCRIPTION:
Smokers of both non-menthol and menthol combustible cigarettes (CC) will be recruited into this AL study to evaluate elements of AL of four heated tobacco products (HTP) (hereinafter, HTP investigational products [IPs]) compared to combustible cigarette (CC) and nicotine polacrilex gum.

Potential subjects may complete a pre-screening telephone interview. They will complete a Screening Visit to assess their eligibility within 45 days prior to check-in (inclusive of enrollment/randomization) and to determine their assignment to either Study Arm 1 (non-menthol smokers) or Study Arm 2 (menthol smokers). Enrollment and clinical conduct for each of the two Study Arms will occur sequentially.

Starting on Day 1, subjects will check-in at the study site to complete procedures to confirm eligibility. Eligible subjects will be enrolled into the appropriate Study Arm and confined for either 11 days (Study Arm 1) or 13 days (Study Arm 2). Based on their Study Arm assignment, subjects will be randomized to a product use sequence (using a Williams Design) in which they will evaluate one IP in each Test Session, including both a high-AL comparator (subject's usual brand [UB] cigarette) and a low-AL comparator (a commercially available nicotine replacement therapy [NRT] nicotine gum). In addition to the AL-comparators, Study Arm 1 will evaluate three HTP IPs (i.e., 5 Test Sessions) and Study Arm 2 will evaluate four HTP IPs (i.e., 6 Test Sessions).

On Day 1 and continuing through Day 11 (Study Arm 1) or Day 13 (Study Arm 2), subjects will participate in Test Sessions that will last for approximately 4 hours. Each Test Session will include collection of both PD measures (subjective and physiological) and PK measures prior to, during and following IP use.

There will be a 1.5-day Product Acclimation Period prior to each Test Session. During the Product Acclimation Period, subjects will be permitted ad libitum use of randomized IP for familiarization prior to use in the next Test Session, as well as ad libitum smoking of their UB cigarettes.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy males or females, 21 to 60 years of age, inclusive, at the time of consent.
3. Smokes combustible, filtered, non-menthol or menthol cigarettes, 83 mm to 100 mm in length. Smokers that also use other tobacco products (e.g., ENDS, smokeless tobacco, heated tobacco products) will not be excluded from study participation.
4. Smokes an average of at least 10 cigarettes per day (CPD) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the PI.
5. Agrees to smoke the same UB cigarette throughout the study period. The UB cigarette is defined as the reported cigarette brand style currently smoked most frequently by the subject.
6. Expired breath carbon monoxide (ECO) level is ≥ 10 ppm and ≤ 100 ppm at Screening and at check-in Day 1.
7. Positive urine cotinine test at Screening.
8. Response at Screening to the Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes".
9. Willing to use UB cigarette, HTP IPs, and Nicorette nicotine gum during the study period.
10. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to the start of each Test Session (either 5 or 6 sessions depending on the Study Arm).
11. Females must be willing to use a form of contraception acceptable to the PI from the time of signing the informed consent until End-of-Study.
12. Agrees to an in-clinic confinement of 11 days (10 nights) for Study Arm 1 -or- 13 days (12 nights) for Study Arm 2.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
4. History or presence of bleeding or clotting disorders.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
6. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes at Screening and at check-in Day 1.
7. Weight of ≤ 110 pounds.
8. Hemoglobin level is < 12.5 g/dL for females or < 13.0 for males g/dL at Screening.
9. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
10. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or check-in Day 1.
11. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
12. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to signing the ICF.
13. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or self-reports a previous attempt within (≤) 30 days prior to signing the ICF.
14. Any use of aspirin (≥ 325 mg/day) or anticoagulants.
15. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
16. Whole blood donation within 8 weeks (≤ 56 days) prior to signing the ICF. NOTE: Subjects will be advised against scheduling a whole blood donation for at least 7 days following study completion.
17. Plasma donation within (≤) 7 days prior to signing the ICF. NOTE: Subjects will be advised against scheduling a plasma donation for at least 7 days following study completion.
18. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
19. Participation in another clinical trial within (≤) 30 days prior to signing the informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
20. Drinks more than 21 servings of alcoholic beverages per week.
21. Has a positive alcohol result at Screening or check-in Day 1.
22. Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
AUECPL 5-240 | 5 minutes to 240 minutes
  area-under-the-effects curve (AUEC) for PL numeric rating scale (NRS) score-versus-time curve from 5 minutes to 240 minutes after the start of IP use.
Emax PL | 240 minutes
  maximum product liking (PL) numeric rating scale (NRS) score after the start of IP use.

CONTACTS AND LOCATIONS:
Overall Officials: Milly Kanobe, PhD, Study Director — RAIS
Locations (1):
- AMR Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kanobe MN, Makena P, Prevette K, Baxter SA. Assessment of Abuse Liability and Nicotine Pharmacokinetics of glo Heated Tobacco Products in a Randomized, Crossover Study. Eur J Drug Metab Pharmacokinet. 2024 Nov;49(6):733-750. doi: 10.1007/s13318-024-00921-4. Epub 2024 Oct 25. PMID 39453550